CLINICAL TRIAL: NCT00501501
Title: The Association Between Delivery Method and Maternal Rehospitalization
Status: Completed | Type: Observational
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Other Study IDs: 5
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Last update posted 2007-07-16 (Estimated); Status verified 2007-07

CONDITIONS: Hospitalization
Keywords: Rehospitalization; Cesarean; Vaginal delivery
MeSH Terms: interventions — Cesarean Section

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Cesarean section
Procedure: Vaginal delivery

SUMMARY:
Hypothesis: The rates of rehospitalization after cesarean section are significantly higher than those following spontaneous vaginal delivery and are due mainly to late bleeding and less to infection.

DETAILED DESCRIPTION:
To determine if there is an association between delivery method and maternal rehospitalization rate, the type of association and the reasons for rehospitalization.

The study population will consist women who were rehospitalized in the Western Galilee Hospital following cesarean section and after a vaginal delivery. Demographic data and hospitalization characteristics will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Parturients rehospitalized after delivery

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 1999-01; Study Completion 2000-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ido Solt, MD, Principal Investigator — Western Galilee Hospital
Locations (1):
- Western Galilee Hospital, Nahariya, Israel